CLINICAL TRIAL: NCT01741311
Title: Secondary HIV Prevention and Adherence Among HIV-infected Drug Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Yale University (Other); APT Foundation, Inc. (Other)
Responsible Party: Principal Investigator, Michael Copenhaver, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H12-050; R01DA032290 (NIH)
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Risk Behavior; Medication Adherence; HIV
Keywords: viral load; HIV; CD4; methadone maintenance; substance use; Antiretroviral therapy (ART)
MeSH Terms: conditions — Risk-Taking; Medication Adherence; Substance-Related Disorders | interventions — Holistic Health; Seroconversion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3H+ Group (Experimental): 3H+ (Holistic for HIV) group patients will receive the standard of drug treatment care (i.e., methadone maintenance treatment and case management) plus four weekly 60-minute HIV risk reduction groups, and a 60-minute booster session at 12 weeks, led by two facilitators trained and supervised by a licensed clinical psychologist. 3H+ is an HIV risk reduction and ART adherence intervention that provides coping skills training and is delivered in a group modality, addressing high risk drug- and sex-related HIV risk behaviors and ART adherence for opioid-dependent individuals living with HIV.
  Interventions: Behavioral: 3H+ (Holistic Health for HIV)
- HHRP+ Group (Active Comparator): HHRP+ (Holistic Health Recovery Program) is comprised of 12 two-hour weekly manual-guided group sessions with comprehensive HIV risk reduction content that addresses the medical, emotional, and spiritual needs of opioid-dependent individuals living with HIV. Each session is designed to last 2 hours and is co-facilitated by two trained facilitators, who address potential motivational conflicts of HIV+ individuals by providing them with self-protective as well as altruistic reasons for examining and changing their HIV risk behaviors and improving adherence behavior. Material is presented using cognitive remediation strategies.
  Interventions: Behavioral: HHRP+ (Holistic Health Recovery Program)

INTERVENTIONS:
Behavioral: 3H+ (Holistic Health for HIV) — Four weekly HIV-risk reduction groups and an additional booster group held at week twelve summarizing the previous sessions' content, designed for opioid-dependent individuals living with HIV.
  Arms: 3H+ Group
Behavioral: HHRP+ (Holistic Health Recovery Program) — 12 two-hour group sessions addressing HIV risk reduction behavior and recovery for opioid-dependent individuals living with HIV.
  Arms: HHRP+ Group

SUMMARY:
This study will test whether 3H+ (Holistic Health for HIV) is comparable to the original HHRP+ (Holistic Health Recovery Program) in reducing HIV risk behaviors and improving ART (Antiretroviral Therapy) adherence in a randomized controlled comparative effectiveness trial among 256 HIV+ persons in drug treatment who report unsafe injection drug use practices or sexual risk behavior.

DETAILED DESCRIPTION:
HIV-infected drug users (DUs) remain a target population as they represent a significant vector for the transmission of new HIV infections (Avants et al., 2004; Margolin et al., 2003), which occur through preventable drug- and sex-related HIV risk behaviors. Though numerous evidence-based HIV risk reduction interventions are now widely available as complete intervention packages, few evidence-based interventions have been designed for implementation within common drug treatment community-based organizations (CBOs), such as methadone maintenance programs (MMPs), where many high-risk HIV-infected drug users seek treatment. Moreover, the few evidence-based interventions that are applicable to drug treatment CBOs are not designed to be "community-friendly" and, hence, are unlikely to be implemented as intended or durable within these critical settings.

The investigators have developed a significantly shortened version of the comprehensive evidence-based Holistic Health Recovery Program (HHRP; Avants et al., 2004; Margolin et al., 2003). This shortened version, Holistic Health for HIV (3H+), has demonstrated feasibility and acceptability as well as preliminary evidence of effectiveness in an uncontrolled study within a resource-limited drug treatment CBO. Therefore, this randomized controlled comparative effectiveness trial (RCT) will test the efficacy and cost-effectiveness of 3H+ versus the original gold standard evidence-based intervention(EBI), Holistic Health Recovery Program for HIV+s (HHRP+), targeting HIV+ drug users (DUs).

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* Opioid dependent and enrolled in methadone maintenance treatment
* Report drug- or sex-related HIV risk behavior in previous 6 months
* Able to read and understand the questionnaires, the Audio Computer Assisted Self Interview (ACASI), and consent form
* Available for the full duration of the study with no anticipated circumstances impeding participation
* Not actively suicidal, homicidal, or psychotic as assessed by trained research staff under the supervision of the PI who is a licensed clinical psychologist in Connecticut.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Copenhaver, Ph.D., Principal Investigator — University of Connecticut
Locations (1):
- APT Foundation, New Haven, Connecticut, United States

REFERENCES:
- [Background] Avants SK, Margolin A, Usubiaga MH, Doebrick C. Targeting HIV-related outcomes with intravenous drug users maintained on methadone: a randomized clinical trial of a harm reduction group therapy. J Subst Abuse Treat. 2004 Mar;26(2):67-78. doi: 10.1016/S0740-5472(03)00159-4. PMID 15050083
- [Background] Margolin A, Avants SK, Warburton LA, Hawkins KA, Shi J. A randomized clinical trial of a manual-guided risk reduction intervention for HIV-positive injection drug users. Health Psychol. 2003 Mar;22(2):223-8. PMID 12683743
- See also: University of Connecticut Center for Health, Intervention, and Prevention (CHIP) — http://www.chip.uconn.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Holistic Health for HIV (3H+): Holistic Health for HIV (experimental intervention)
- Holistic Health Recovery Program (HHRP+): Holistic Health Recovery Program (comparison condition in this non-inferiority trial)
Period: Overall Study
Arm/Group | Holistic Health for HIV (3H+) | Holistic Health Recovery Program (HHRP+)
Started | 52 | 54
Completed | 32 | 18
Not Completed | 20 | 36

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3H+ Group | HHRP+ Group | Total
Number analyzed (Participants) | 52 | 54 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 54 | 106
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 30 | 33 | 63
Region of Enrollment [Number; unit: participants]
  United States | 52 | 54 | 106
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 15 | 41
  White | 11 | 22 | 33
  More than one race | 15 | 17 | 32
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 17 | 31
  Not Hispanic or Latino | 37 | 37 | 74
  Unknown or Not Reported | 1 | 0 | 1
Anti-retroviral Therapy (ART) Adherence [Count of Participants; unit: Participants] — Number of participants in each condition reporting optimal (>95%) adherence to anti-retroviral medication using the visual analogue scale (VAS). The VAS measures adherence continuously from 0 to 100%, with higher scores meaning a better outcome. A greater number of participants reporting optimal adherence is better.
  Participants | 32 | 33 | 65

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Each Condition With Optimal ART Adherence
Description: Anti-retroviral therapy (ART) adherence was assessed by self-report using the visual analogue scale (VAS). The VAS measures adherence continuously from 0 to 100%, with higher scores indicating better adherence to the medication. A greater number of participants with optimal ART adherence is better. Optimal ART adherence is defined as a score >95% on the visual analog scale (VAS).
Time Frame: Assessed at post-intervention, 3-months, & 6-months. Reported in the table at 6-months.
Measure: Number; unit: participants
Arm/Group | 3H+ Group | HHRP+ Group
Number analyzed (Participants) | 52 | 54
participants | 27 (0.063) | 29 (0.066)

2. Secondary Outcome: Viral Suppression
Description: Number of participants in each condition with viral load suppression at the 6-month assessment point. Viral suppression (VS) is defined as someone having HIV-1 RNA<50 copies/mL. A greater number of participants with VL suppression is a better outcome.
Time Frame: Assessed at post-intervention, 3-months, & 6-months. Reported in the table at 6-months.
Measure: Count of Participants; unit: Participants
Groups:
- Holistic Health for HIV (3H+): 3H+
- Holistic Health Recovery Program (HHRP+): HHRP+
Arm/Group | Holistic Health for HIV (3H+) | Holistic Health Recovery Program (HHRP+)
Number analyzed (Participants) | 52 | 54
Participants | 45 (0.048) | 34 (0.066)

ADVERSE EVENTS:
Time Frame: Adverse event collection occurred starting at baseline, and then continued at post-intervention,and then at the 3 month and 6-month follow-up points.
Groups:
- Holistic Health for HIV (3H+): Holistic Health for HIV (experimental condition in this non-inferiority trial) - This is an adapted/abbreviated version of the comprehensive evidence-based gold standard.behavioral HIV risk reduction approach that is designed for HIV-infected opioid-dependent persons enrolled in drug treatment
- HHRP+: Holistic Health Recovery Program (gold standard evidence-based comparison condition in this non-inferiority trial) that was designed for HIV-infected opioid-dependent persons enrolled in drug treatment.
Arm/Group | Holistic Health for HIV (3H+) | HHRP+
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/54
Other Adverse Events (participants affected / at risk) | 0/52 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-07-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT01741311/Prot_SAP_000.pdf